CLINICAL TRIAL: NCT04951154
Title: Collection of Peripheral Blood and Lung Lesion Samples From Participants With Suspected Lung Cancer to Examine the Potential of Bronchoscopic Biopsies to Assess Non-small Cell Lung Cancer (NSCLC) Tumor Immune Subtypes and Related Biomarkers
Brief Title: A Study to Examine Biomarkers From Lung and Blood Samples in Participants With Suspected Lung Cancer
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109030; NOPRODLUC0002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-07-01; First posted 2021-07-06 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Suspected Lung Cancer: Eligible participants with suspected lung cancer will be enrolled and undergo diagnostic and research bronchoscopic biopsies and research blood sample collection for biomarker analysis. Those participants who proceed to surgical resection will have additional research samples taken from the resected tumor and additional research blood samples drawn for biomarker analyses at the resection visit and at the post-operative follow up visit. Participants will then be followed clinically for two years for evidence of recurrence or until participants with confirmed lung cancer recurrence, whichever occurs earlier.
  Interventions: Other: Bronchoscopic Biopsy; Other: Blood Sample

INTERVENTIONS:
Other: Bronchoscopic Biopsy — Bronchoscopic biopsies will be used to evaluate biomarkers of tumor biology and immunology.
  Other Names: No investigational product will be administered in this study.
Other: Blood Sample — Blood samples will be obtained to measure circulating biomarkers.
  Other Names: No investigational product will be administered in this study.

SUMMARY:
The purpose of this study is to assess spontaneous residual viable tumor cells (RVT) in the surgically resected tumor (Non-small cell lung cancer [NSCLC]).

DETAILED DESCRIPTION:
This is a multicenter study including participants with a radiographically identified lung lesion that is highly suspicious for lung cancer that has been deemed likely to be resectable. After confirmation of a NSCLC diagnosis and eligibility for surgical resection with curative intent, participants will undergo surgical resection of their tumor. Participants will complete a follow up visit approximately 2-4 weeks after their surgery. During this initial period of the study, blood and tissue samples will be collected for biomarker analyses. Participants will then receive a follow up telephone call every 6 months for up to an additional 2 years, or until participants with confirmed lung cancer recurrence, whichever occurs earlier, to document any instances of disease recurrence. Therefore, a key objective of this study is to achieve a more detailed understanding of how representative these pretreatment bronchoscopic biopsies are of the resected tumor sample, hence, no investigational new treatments will be given to the participants enrolled in this study. Safety will be evaluated by monitoring of procedure-related adverse events (AEs) and serious adverse events (SAEs). The total duration of the study will be approximately 2 years and 3 months (actual duration of participation will be dependent upon timing of scheduling of bronchoscopy and surgical resection and timing of cancer recurrence, if applicable).

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more radiographically identified 1-5 centimeter (cm) solid or sub-solid lung lesions with at least a 1 cm solid component highly suspicious for lung cancer and requiring bronchoscopic diagnosis, with a computed tomography (CT) scan or other cross-sectional imaging (example, CT-positron emission tomography [PET]) within 28 days of the intended bronchoscopy
* Deemed by the investigator(s), including thoracic surgeon, to be a suitable candidate for surgical resection with curative intent, following review of participant information which may include past medical history, medications, pulmonary function testing, and CT scan
* Able to tolerate general anesthesia and a diagnostic bronchoscopy, as assessed by the investigator
* Each participant (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of the study and the procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Participants who are currently receiving, have received within the last 6 months, or plan to receive any systemic treatment for their presumed lung cancer between Screening visit and the last blood sample collection at Week 6 visit
* Participants who have previously received radiation therapy to the lung (example, radiation therapy to chest wall, such as for breast cancer is allowed)
* Participants who are currently receiving systemic steroids or other immunosuppressive medications (example, methotrexate, azathioprine, anti- tumor necrosis factor [TNF] agents), have received these medications within 6 weeks prior to bronchoscopic biopsy, or who plan to receive these medications between Screening visit and last blood sample collection at Week 6 visit. Periprocedural low dose systemic steroids may be given during bronchoscopy and surgical resection procedures per institutional standard of care (SOC) but cannot be administered before blood samples have been collected. Use of inhaled or other topical corticosteroids (example, otic, ocular, skin) is permitted
* Participants with uncorrectable coagulopathy (example, hemophilia, disseminated intravascular coagulation [DIC], massive pulmonary embolism [PE]) or with therapeutic anticoagulant that cannot be held for an appropriate interval prior to the procedure
* Any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise the well-being) or physical limitations that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants with a radiographically identified lung lesion that is highly suspicious for lung cancer that has been deemed likely to be resectable.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Percent of Residual Viable Tumor Cells (% RVT) at the Time of Non-small Cell Lung Cancer (NSCLC) Resection | Up to Week 6
  Percent of RVT cells at the time of NSCLC resection will be reported.

SECONDARY OUTCOMES:
Tumor Gene Expression Analysis by Ribonucleic Acid (RNA)-sequencing or Polymerase Chain Reaction (PCR) Techniques | Up to 6 Weeks
  RNA sequencing or PCR techniques will be used to assess tumor gene expression.
Tumor Mutational Burden Assessed by Next Generation Sequencing | Up to 6 Weeks
  Sequencing nucleic acids by next generation sequencing will be used to calculate tumor mutational burden.
Tissue Frequencies of Immune Cell Subsets Determined via Semi-quantitative Immunofluorescence and/or Imaging Mass Cytometry | Up to 6 Weeks
  Percentage of immune cell subsets measured using immunofluorescence and/or imaging mass cytometry will be reported.
T-cell Receptor (TCR) Repertoire Sequencing in Tumor | Up to 6 Weeks
  T cell receptor (TCR) sequencing in tumor samples will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- United States (2):
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No